The Influence of

Postoperative Analgesia

on Systemic Inflammatory

Response and POCD

After Femoral Fractures

Surgery

Document Date: May 26, 2017

NCT02848599

ID: 25-1:6563-3/2014

Category data were represented by absolute and relative frequencies. Variations of category variables were tested by Fisher's exact test. The numerical data are described by the median and the limits of the interquartile range. The normality of distribution of observed numeric variables was tested by the Shapiro -Wilk test. The differences between the normal distribution of numeric variables between the two independent groups were tested by Mann-Whitney's In Test. To determine the difference between the two dependent samples, Friedman's test was used. Logistic regression was used to assess the influence of several factors on the likelihood that POCD would develop in the observed subjects. The receiver operating curve (ROC) analysis was used to determine the optimal threshold, area under the curve (AUC), specificity, and sensitivity of the tested parameters. All P values were two-tailed. The level of significance was set at Alpha = 0.05. The statistical analysis was performed using MedCalc Statistical Software version 14.12.0 (MedCalc Software bvba, Ostend, Belgium; http://www.medcalc.org; 2014)